CLINICAL TRIAL: NCT04539210
Title: Completely Edentulous Patients Screw-retained Maxillary Complete Denture With Electric Welded Metal Framework Versus Cast One, Patient Satisfaction Assessment (Randomized Control, Split Mouth Trial)
Brief Title: Screw-retained Maxillary Complete Denture With Electric Welded Metal Framework Versus Cast One, Patient Satisfaction Assessment.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, fatma hussein abd elmonem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO6-2-1
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-04

CONDITIONS: Patient Satisfaction; Maintenance
Keywords: electric welding; metal framework
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric Welded Metal Framework (Experimental): A preexisting or prepared flat surface area of the welding abutment of implant at central incisor position at one side (right or left) will serve as the welding point. A titanium bar will be shaped following the curvature of the implants positioned. At this point, temporary titanium implant abutments will be welded with the titanium bar in the oral cavity, using the Syncrystallization Unit. Finally, the prosthetic framework, created by welding the titanium bar to the implant abutments, will be removed and opaque will be applied in order to avoid metal shining through the acrylic resin. The framework is picked up to denture with hard liner, and screwed to the denture.
  Interventions: Device: Electric Welded Metal Framework
- cast metal framework (Experimental): On a verified analogue model, occlusion blocks will be constructed for adjustment of vertical dimension and bite registration. Afterwards, CCM abutments will be fastened over the analogues of the placed implants, followed by waxing, spruing and casting. The resultant cast metal framework will be inserted inside the patient's mouth on the right or left installed implants to insure passivity of fit. In case of framework misfit, separation will be performed using a disc, followed by intraoral splinting and soldering. After framework soldering, another try-in will be done to insure framework fit.
  Interventions: Device: Electric Welded Metal Framework

INTERVENTIONS:
Device: Electric Welded Metal Framework — Screw-retained Maxillary Complete Denture With Electric Welded Metal Framework

SUMMARY:
In this study the investigators are going to compare the effect of electric welded metal frame work and cast frame work on patient satisfaction and maintenance of the final prosthesis.

DETAILED DESCRIPTION:
In this study twelve completely edentulous patients will be enrolled and In each patient six implants will be inserted in the maxillary arch at crestal bone level in predefined positions (positions 15, 13, 11, 21, 23, 25) with the help of a surgical template following a submerged healing protocol and checked for primary stability clinically. After a 4-month osseointegration period, second-stage surgery will be performed and healing abutments will be placed. After the second-stage surgery, prosthetic procedures will be initiated.

then for one side (the intervention side) the metal framework will be constructed as follow: A preexisting or prepared flat surface area of the welding abutment of implant at central incisor position at one side (right or left) will serve as the welding point. A titanium bar will be shaped following the curvature of the implants positioned. At this point, temporary titanium implant abutments will be welded with the titanium bar in the oral cavity, using the Syncrystallization Unit .The welding process is electrical and protected by an argon gas supply (Syncrystallization). The equipment allows the welding of metallic elements directly in the mouth. Current flowing through the contact points, being in contact with the parts to weld, warms up to the point of fusion, achieving a solid, welded junction. Then will be placed between the two electrodes of a welding clamp. The energy contained in a previously unloaded battery of capacitors is transferred to the electrodes of the welding cycle is subdivided in three stages: Pre-gas, welding, and post-gas phase. While the pre-gas phase allows an oxygen-free welding point prior to the actual fusion, the post-gas phase ensures the absence of oxygen and subsequent oxidation during cooling. Finally, the prosthetic framework, created by welding the titanium bar to the implant abutments, will be removed and opaque will be applied in order to avoid metal shining through the acrylic resin.

for the other side :

At the day of second stage surgery restoration will be fabricated as follow:

For the cast metal framework group, CCM abutments (Titanium base abutments with a plastic cast able sleeve) will be fastened over the analogues of the placed implants, on a verified analogue model.

For the preparation of the verified model, open tray (pick-up) impression copings will be fastened to the placed implants, and an un splinted impression will be made using addition silicone impression material in a single step manner, using putty and light consistency addition silicone.

A stone model will be obtained after fastening of the implant analogues, fabrication of a gingival mask and pouring the impression using extra-hard dental stone. Over the obtained stone model, splinting of the open tray impression copings will be performed using duralay resin to obtain a jig that will be further separated and resplinted intra orally, over which a splinted pick-up impression will be remade. The new impression will be poured into extra-hard stone after fabricating a gingival mask.

On the verified master analogue model, occlusion blocks will be constructed for adjustment of vertical dimension and bite registration. Afterwards, CCM abutments will be fastened, followed by waxing, spruing and casting. The resultant framework will be inserted inside the patient's mouth on the following implants; right or left implants installed; central, canine, and second premolar to insure passivity of fit. In case of framework misfit, separation will be performed using a disc, followed by intraoral splinting using duralay resin and soldering. After framework soldering, another try-in will be done to insure framework fit, then the final pick-up of the framework into the denture will be performed. Then the final prosthesis will be sectioned at the midline resulting two separate super structures.

then Patient satisfaction will be assessed using Boerrigter's method questionnaire after 3,6 and 12 months.

During the 12 months follow-up period as follow(within 2weaks of delivery,6months after delivery and 12 months after delivery) , number of prosthodontic complications for the laser welded and cast metal framework supported over dentures will be registered and calculated according to the following events: screw loosening of the abutment, screw loosening of the prosthesis, fracture of the screw of the abutment, fracture of the screw of the prosthesis, abutment fracture, framework fracture, fracture of acrylic resin denture, loss of cover of access hole, prosthetic teeth fracture and remake of the prosthesis, occlusal discrepancies ,maxillary and mandibular denture relining if needed ,pain.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 45 to 65 years old.
* Absence of any medical disorder that could complicate the surgical phase or affect osseointegration .
* The patients must be completely edentulous.
* The patient must have enough bone height for implants, minimum length of bone 10mm and a minimum diameter of bone 5 mm.
* Patients with good oral hygiene.
* Complete denture wearer.
* Adequate inter arch space for screw retained prosthesis.
* Absence of any intra-oral pathological condition.

Exclusion Criteria:

* Patients with recent extraction(less than three months).
* Patients with inflamed ridge or candida infection.
* Patients with flappy ridge.
* Para functional habits.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 12 months
  satisfaction assessed by Boerrigter's method questionnaire.in this questionnaire, there are three aspects to consider:(1) problems with the denture itself;(2) masticating ability; and (3) overall denture performance. different answers to each question are assigned scores and the total score can be calculated for further evaluation and analysis.

SECONDARY OUTCOMES:
Maintenance of the final prosthesis | 12 months
  During the 12 months follow-up period as follow(within 2weaks of delivery,6months after delivery and 12 months after delivery) , number of prosthodontic complications for the laser welded and cast metal framework supported over dentures will be registered and calculated according to the following events: screw loosening of the abutment, screw loosening of the prosthesis, fracture of the screw of the abutment, fracture of the screw of the prosthesis, abutment fracture, framework fracture, fracture of acrylic resin denture, loss of cover of access hole, prosthetic teeth fracture and remake of the prosthesis, occlusal discrepancies ,maxillary and mandibular denture relining if needed ,pain.

CONTACTS AND LOCATIONS:
Overall Officials: cairo university, Study Director — cu
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No